CLINICAL TRIAL: NCT01351376
Title: The Effectiveness of Low Level Laser Therapy (LLLT)Combined With Complex Decongestive Therapy (CDT) in the Treatment of Breast Cancer-Related Lymphedema: A Double-Blind, Randomized, Placebo-Controlled Study
Brief Title: LLLT Combined With CDT in Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-00923
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Lymphedema, Low Level Laser, Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Placebo (Placebo Comparator): CDT + inactive LLL
  Interventions: Device: Low Level Laser Therapy
- LLL combined with CDT (Active Comparator): CDT + active LLL
  Interventions: Device: Low Level Laser

INTERVENTIONS:
Device: Low Level Laser Therapy — Placebo LLL combined with CDT
  Other Names: Low Level Laser; Complex Decongestive Therapy
  Arms: Placebo
Device: Low Level Laser — Active LLL combined with CDT
  Other Names: Complex Decongestive Therapy
  Arms: LLL combined with CDT

SUMMARY:
This study aims to explore the effects of Low Level Laser Therapy (LLLT) on breast cancer-related lymphedema when utilized in conjunction with Complex Decongestive Therapy (CDT) when compared to CDT treatment alone. The investigators hypothesize that the addition of LLLT to CDT will result in statistically significant improvements and greater long-term benefits as measured by changes in arm volume and quality of life when compared to the benefits of CDT alone for the treatment of breast cancer-related lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* unilateral breast cancer with ipsilateral lumpectomy or mastectomy and lymph node dissection (sentinel biopsy or axillary dissection)
* stage II or III unilateral secondary upper extremity lymphedema (as defined by the International Society of Lymphology)
* girth ≥ 2 cm circumferential difference and/or volume ≥ 200 mL compared to the uninvolved upper extremity at any 4 cm segment
* able to commit to a long term follow-up schedule

Exclusion Criteria:

* active cancer/metastatic cancer
* currently receiving or have plans for adjuvant radiation or chemotherapy
* pregnant
* presence of other extremity lymphedema (primary or secondary)
* pacemaker
* artificial joints in the upper quadrants
* renal failure
* arterial insufficiency
* congestive heart failure
* chronic inflammatory conditions
* history of deep vein thrombosis (DVT) in the lymphedematous upper extremity
* previous treatment with Low Level Laser (regardless of indication)
* medication(s) known to affect body fluid balance
* body mass index (BMI) > 40 (morbid obesity)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Denham, PT, MA, Principal Investigator — NYU Rusk Institute of Rehabilitation Medicine
Locations (3):
- United States (3):
  - NYU Clinical Cancer Center, New York, New York
  - NYU Rusk Institute of Rehabilitation Medicine, New York, New York
  - Tisch Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | LLL Combined With CDT
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LLL Combined With CDT | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Arm Volume
Time Frame: 13 Months
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Placebo | LLL Combined With CDT
Number analyzed (Participants) | 10 | 11
cm^3 | 1.48 (1.01) | 1.58 (1.0)

2. Secondary Outcome: Short-Form Health Survey (SF-36)
Description: Short Form Health Survey (SF-36), an instrument composed by 8 subscales: Physical Functioning, Physical Role Function, Bodily Pain, General Health, Vitality, Social Functioning, Emotional Role Function and Mental Health. The individual question items (Likert scale 0-4) are first summed for each item under the various sections. Then, those summary scores are then standardized on a scale between 0 and 1 using the mean and standard deviation of the actual scores and finally, weighted to a scale between 0 and 100. The items contributing to a scale are scored so that a higher score represents better health, and they are averaged together to create the scale score. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | LLL Combined With CDT
Number analyzed (Participants) | 10 | 11
score on a scale | 75.5085 (16.07351) | 72.6042 (18.01269)

ADVERSE EVENTS:
Arm/Group | Placebo | LLL Combined With CDT
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No